CLINICAL TRIAL: NCT00002448
Title: Evaluation of Immune Reconstitution in HIV Infected Patients Treated With Fortovase (Saquinavir) SGC QD Plus Ritonavir QD Plus 2 NRTIs Vs Efavirenz QD Plus 2 NRTIs
Brief Title: A Study to Compare the Effects of Two Anti-HIV Drug Combinations on the Immune Systems of HIV-Infected Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Model: Parallel | Purpose: Treatment
Other Study IDs: 229S; M61028
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-01

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; HIV Protease Inhibitors; Ritonavir; Dosage Forms; Saquinavir; Reverse Transcriptase Inhibitors; Anti-HIV Agents; efavirenz
MeSH Terms: conditions — HIV Infections | interventions — Ritonavir; efavirenz; Saquinavir

INTERVENTIONS:
Drug: Ritonavir
Drug: Efavirenz
Drug: Saquinavir

SUMMARY:
The purpose of this study is to examine how the immune systems of HIV-infected patients react to 2 anti-HIV drug combinations.

DETAILED DESCRIPTION:
Patients are randomized to two study arms for at least 48 weeks of treatment. Arm A receives SQV SGC plus RTV plus two NRTIs of choice. Arm B receives EFV plus two NRTIs of choice. NRTIs approved for study use are stavudine (d4T), didanosine (ddI), zidovudine (AZT), lamivudine (3TC), Combivir, and zalcitabine (ddC). Abacavir is excluded. The following immunology variables and HIV-1 viral characteristics will be evaluated during study visits: CD4 and CD8 cell counts; naive and memory T-cells; T-cell activation markers (HLA-DR and CD38); T-cells expressing T helper 1- (TH1-) and T helper 2- (TH2-) associated intracytoplasmic cytokines; anti-CD3 T-cell activation responses; T-cell receptor V Beta repertoire; cytotoxic T-lymphocyte (CTL) activity levels; lymph node histology (optional); HIV-1 qualitative microcultures and viral phenotyping for non-syncytium-inducing (NSI) and syncytium-inducing (SI) viral isolates. Laboratory determinations, adverse effects, neurological exams (including mental status evaluations), and lipodystrophy parameters (including fasting lipid profile and physical parameters) also are evaluated.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are HIV-positive.
* Have a viral load of at least 5,000 copies/ml and a CD4 cell count greater than 75 cells/mm3.
* Are at least 16 (need consent of parent or guardian if under 18).
* Are able to complete the study.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Have ever taken anti-HIV medications.
* Are pregnant or breast-feeding.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40
Dates: Start 1999-10

CONTACTS AND LOCATIONS:
Overall Officials: Mark Holodniy, Principal Investigator; Joseph John, Study Chair; Ronald Mitsuyasu, Study Chair
Locations (3):
- United States (3):
  - UCLA Care Ctr, Los Angeles, California
  - Palo Alto Veterans Affairs Health Care System, Palo Alto, California
  - Robert Wood Johnson Med School/UMDNJ, New Brunswick, New Jersey